CLINICAL TRIAL: NCT05321732
Title: A Randomized, Open-label, Multiple-dose, Crossover Clinical Trial to Investigate the Drug Interaction of DWP16001 and DWC202010 After Oral Administration in Healthy Adults
Brief Title: The Drug Interaction of DWP16001 and DWC202010 After Oral Administration in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP306001101
Record Dates: First submitted 2022-01-16; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Enavogliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention: DWP16001 A mg (Experimental)
  Interventions: Drug: DWP16001
- Intervention: DWC202010 B mg (Experimental)
  Interventions: Drug: DWP202010
- Intervention: DWP16001 A mg + DWC202010 B mg (Experimental)
  Interventions: Drug: DWP16001; Drug: DWP202010

INTERVENTIONS:
Drug: DWP16001 — DWP16001 A mg
  Arms: Intervention: DWP16001 A mg; Intervention: DWP16001 A mg + DWC202010 B mg
Drug: DWP202010 — DWP202010 B mg
  Arms: Intervention: DWC202010 B mg; Intervention: DWP16001 A mg + DWC202010 B mg

SUMMARY:
This study aims to evaluate the pharmacokinetic and pharmacodynamic characteristics and safety of co-administration of DWP16001 2 mg and DWC202010 (DWC202010 37.5 mg) in healthy adults compared to the case of administration alone.

DETAILED DESCRIPTION:
The study design is a randomized, open-label, multiple-dose, crossover clinical trial. The patients were randomly assigned to each group. Primary endpoint was Cmax,ss and AUCtau,ss of DWP16001 and DWC202010. Secondary endpoints were Cmax,ss, Tmax,ss, t1/2, CLss/F, fluctuation of DWP16001 and DWC202010, and Cmax,ss, Cmin,ss, AUCtau,ss, Tmax,ss, and metabolic ratio of DWP16001 metabolites(M1).

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax,ss) of DWP16001 | Before IP administration of Day 1, Day 5, and Day 6
Area under the plasma concentration versus time curve (AUCtau,ss) of DWP16001 | Before IP administration of Day 1, Day 5, and Day 6
Peak Plasma Concentration (Cmax,ss) of DWC202010 | Before IP administration and post-dose up to 24 hours
Area under the plasma concentration versus time curve (AUCtau,ss) of DWC202010 | Before IP administration and post-dose up to 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Yoon S, Park MS, Jin BH, Shin H, Na J, Huh W, Kim CO. Pharmacokinetic and pharmacodynamic interaction of DWP16001, a sodium-glucose cotransporter-2 inhibitor, with phentermine in healthy subjects. Expert Opin Drug Metab Toxicol. 2023 Jul-Dec;19(7):479-485. doi: 10.1080/17425255.2023.2249397. Epub 2023 Aug 25. PMID 37593838